CLINICAL TRIAL: NCT01537250
Title: A Multi-center, Randomized, Double-blind, Double-dummy Parallel-controlled Phase II Clinical Study to Assess the Efficacy and Safety of Nemonoxacin Malate in Treating Adult Patients With Community-acquired Pneumonia (CAP)
Brief Title: Phase II Clinical Study to Assess the Efficacy and Safety of Nemonoxacin Malate in Treating Adult Patients With Community-acquired Pneumonia (CAP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TaiGen Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TG-873870-C-3
Record Dates: First submitted 2012-02-05; First posted 2012-02-23 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Community-acquired Pneumonia
Keywords: CAP
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Levofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nemonoxacin 750 mg (Active Comparator): Nemonoxacin 750 mg 2 tablets.
  Interventions: Drug: Levofloxacin 500 mg placebol
- Nemonoxacin 500 mg (Active Comparator): Nemonoxacin 500 mg 3 tablets
  Interventions: Drug: Levofloxacin 500 mg placebol
- Levofloxacin 500 mg (Active Comparator): Levofloxacin 500 mg
  Interventions: Drug: Nemonoxacin 3 tablets

INTERVENTIONS:
Drug: Levofloxacin 500 mg placebol — oral form,,once adily,7~10 days
  Arms: Nemonoxacin 750 mg
Drug: Levofloxacin 500 mg placebol — oral form,,once adily,7~10 days
  Arms: Nemonoxacin 500 mg
Drug: Nemonoxacin 3 tablets — oral form,once daily,7~10 days
  Arms: Levofloxacin 500 mg

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and population pharmacokinetics of oral nemonoxacin in community-acquired pneumonia (CAP) subjects.

DETAILED DESCRIPTION:
Evaluate clinical efficacy, microbiological efficacy and safety of Nemonoxacin adult patients with community-acquired pneumonia (CAP); and

A study on the population pharmacokinetics (PPK) of continuous oral administration of Nemonoxacin in adult patients with CAP.

ELIGIBILITY:
Inclusion Criteria:

1. age of 18~70, BMI ≥ 18 kg/m2
2. Female patients must avoid pregnancy
3. Patients who are clinically diagnosed with community-acquired pneumonia (CAP)
4. Chest X-ray shows inflammatory exudation or infiltration image.
5. Patients who used antibacterial agents (excluding quinolones) within 72 hours before
6. The patient's disease condition permits oral administration

Exclusion Criteria:

1. Patients who have any of bronchiectasis and pulmonary disease.
2. Hospitalized within 14 days before enrollment
3. Have a history of allergy to any quinolone or fluoroquinolone antibiotic
4. Patients who suffered uncontrolled mental disorders, epilepsy or central nervous system diseases.
5. Renal, liver insufficiency
6. Malabsorption syndrome or other gastrointestinal diseases
7. Immune system diseases,such as a history of human immunodeficiency virus (HIV) infection,neutropenia or malignant tumor in the blood system or a solid organ, or removal of spleen
8. Steroids longterm use, the dose is at least 20mg of prednisone daily
9. Patients under critical condition.
10. Shows significant abnormality of the cardiac conduction system (CCS) or other abnormalities, or prolonged QTc
11. Have a medical history of prolonged QTc, or require concomitant medication of drugs that will lead to prolongation of QTc
12. Patients who received chemotherapy or anti-tumor therapy within 6 months
13. Alcohol abused or drugs banned
14. Patients who used quinolones within two weeks before enrollment
15. Donated more than 500ml of blood within 3 months
16. co-medication of other antibacterial agents required.
17. by investigators judgement,patient who increase the risk to the subjects or interfere with this clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2009-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Per subject clinical cure rate | 16days
  Clinical cure rate equals to number of clinical evaluable divided by number of clinical cured. If subject's clnical outcome is evaluable by principal invastigator, he/she is defined as clinical evaluable.
Per subject microbiological cure rate | 16days
  Microbiological cure rate equals to number of microbiological evaluable divided by number of eradicated or presumed eradicated.

SECONDARY OUTCOMES:
Pharmacokinetic profile of nemonoxacin in CAP subjects | 3days

CONTACTS AND LOCATIONS:
Overall Officials: Yingyuan Zhang, PhD, Principal Investigator — Huashan Hospital, Fundan University
Locations (32):
- China (32):
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing
  - Beijing Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - PLA Second Artillery General Hospital, Beijing
  - Zhen Hospital, Capital Medical University Beijing, Beijing
  - Daping Hospital, Third Military Medical University, Chongqing
  - First Affiliated Hospital of Fujian Medical University, Fujian
  - Gansu Provincial People's Hospital, Gansu
  - Guangzhou Red Cross Hospital, Guangzhou
  - Second Affiliated Hospital of Sun Yat-sen, Guangzhou
  - Affiliated Hospital of Guilin Medical College, Guilin
  - Taihe Hospital in Shiyan City, Hubei Province, Hubei
  - Third Xiangya Hospital, Central South University, Hunan
  - Jiangxi Provincial People's Hospital, Jiangxi
  - Second Affiliated Hospital of Nanchang University, Jiangxi
  - Jinan Central Hospital, Jinan
  - Shengjing Hospital of China Medical University, Liaoning
  - Nanjing General Hospital of Nanjing Military Region, Nanjing
  - Huashan Hospital ,Fudan University, Shanghai
  - Institute of Antibiotics, Huashan Hospital, Fundan University, Shanghai
  - Institute of Antibiotics,Huashan Hospital ,Fudan University, Shanghai
  - Shanghai Pudong New Area, Oriental Hospital, Shanghai
  - Shanghai Putuo District Central Hospital, Shanghai
  - First Hospital of Shanxi Medical University, Shanxi
  - People's Liberation Army General Hospital of Shenyang Military Region, Shenyang
  - Shenzhen People's Hospital, Shenzhen
  - West China Hospital of Sichuan University (Respiratory), Sichuan
  - Second Affiliated Hospital of Wenzhou Medical College, Wenzhou
  - People's Hospital of Wuhan University, Wuhan
  - Wuhan General Hospital of PLA Guangzhou Military Region, Wuhan
  - First Affiliated Hospital, Zhejiang University School of Medicine, Zhejiang

REFERENCES:
- [Derived] Liu Y, Zhang Y, Wu J, Zhu D, Sun S, Zhao L, Wang X, Liu H, Ren Z, Wang C, Xiu Q, Xiao Z, Cao Z, Cui S, Yang H, Liang Y, Chen P, Lv Y, Hu C, Lv X, Liu S, Kuang J, Li J, Wang D, Chang L. A randomized, double-blind, multicenter Phase II study comparing the efficacy and safety of oral nemonoxacin with oral levofloxacin in the treatment of community-acquired pneumonia. J Microbiol Immunol Infect. 2017 Dec;50(6):811-820. doi: 10.1016/j.jmii.2015.09.005. Epub 2015 Dec 1. PMID 26748734